CLINICAL TRIAL: NCT04974567
Title: Tear Based Sample Collection for Breast Cancer Detection
Brief Title: Tear Based Sample Collection Breast Cancer Detection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Namida Lab (Industry)
Collaborators: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: IRB # 21-0026
Record Dates: First submitted 2021-06-24; First posted 2021-07-23 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Tear; Breast Cancer Female
Keywords: preventative screening; protein biomarkers; lacrimal tear fluid; mammography; ELISA assay; CLIA laboratory; lab developed test; high complexity; tear collection; mammogram; improved patient outcomes; reduce gap in access; health equity; total cost of care; trust from patient; increased compliance; affordable; low cost; non-invasive; women's health and wellness; breast health; breast cancer screening test
MeSH Terms: conditions — Breast Neoplasms; Lacerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lacrimal (tear) fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women recently diagnosed with breast cancer who have not undergone any treatment.: Tear sample collection
  Interventions: Other: Schirmer Strip

INTERVENTIONS:
Other: Schirmer Strip — A tear-based screening assay for breast cancer developed and validated by Namida Lab, Inc., a high complexity CLIA certified lab. It consists of two parts: tear sample collection using a Schirmer Strip and a clinical lab-developed test that measures protein biomarkers for breast cancer screening.

SUMMARY:
This study aims to collect tear samples from 50 women who have been recently diagnosed with breast cancer.

DETAILED DESCRIPTION:
Namida Lab, Inc. is a biotechnology company located in Fayetteville, AR, with a certified, high-complexity CLIA lab. In January of 2021, Namida Lab, Inc. completed the analytical and clinical validation of a tear-based biological screening test for breast cancer based on proteins from tears. The validation process was carried out manually and now needs to be conducted on the Hamilton StarPlus automated ELISA system. To complete the robot validation, Namida Lab, Inc. needs fifty (50) tear samples collected from women recently diagnosed with breast cancer but who have not undergone any treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individual is an adult woman and has recently been diagnosed with breast cancer.

Exclusion Criteria:

* Individual is excluded if they have already started treatment for the breast cancer diagnosis.
* Age less than 18 or more than 100 years.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Tear Based Breast Cancer Detection study participants are all women, born biologically female, with a recent diagnosis of breast cancer, have not started treatment, and are between the ages of 18 to 100 years old.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of participant tear samples collected. | 90 days
  The purpose of this study is to collect 50 tear samples from women who have been recently diagnosed with breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Klimberg, MD, PhD, Principal Investigator — UTMB Health
Locations (1):
- UTMB Health, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared or made available to other researchers.

DOCUMENTS (2):
  • Study Protocol (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT04974567/Prot_000.pdf
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04974567/ICF_001.pdf